CLINICAL TRIAL: NCT05412875
Title: A Pilot Trial of Electronic Cigarettes in Patients Diagnosed With Cancers of the Head, Neck, and Lung
Brief Title: Pilot Trial of E Cigarettes in Pts Diagnosed With Cancer of the Head, Neck, and Lung
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding lapse
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Theodore Brasky PhD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21255; NCI-2022-00864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K07CA215546 (NIH)
Record Dates: First submitted 2022-05-17; First posted 2022-06-09 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Lung Non-Small Cell Carcinoma; Stage I Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (JUUL) (Experimental): Beginning 1 month before surgery, patients receive a JUUL e-cigarette and a 1 month supply e-liquid pods. After completion of surgery, patients receive another 1 month supply of e-liquid pods.
  Interventions: Drug: Nicotine Replacement; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Given usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Drug: Nicotine Replacement — Given JUUL
  Other Names: Nicotine Replacement Therapy; NRT
  Arms: Arm I (JUUL)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial investigates the acceptability of electronic cigarettes (JUUL) for smoking cessation (quitting smoking) and the reduction of surgery-related complications in patients with newly diagnosed head, neck, or lung cancer. Smoking before surgery is associated with increased risk of complications during and after surgery. Electronic cigarettes are a type of special product that gives small, steady doses of nicotine to help stop cravings and relieve symptoms that occur when a person is trying to quit smoking. Stopping cigarette smoking before surgery may reduce the risk of complications during and after surgery in patients with head, neck, or lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate feasibility, acceptability, compliance, and safety of a non-randomized 2-month trial of a pod based electronic cigarette (intervention) versus usual care for stage I-III lung cancer patients and stage I-IV head and neck cancer patients undergoing surgical resection.

II. Examine the effect of the pod based electronic cigarette (intervention) on surgical complications, quality of life, and whether it promotes complete or incomplete switching to the non-combustible product.

OUTLINE: Patients choose to participate in 1 of 2 arms.

ARM I: Beginning 1 month before surgery, patients receive a JUUL e-cigarette and a 1 month supply e-liquid pods. After completion of surgery, patients receive another 1 month supply of e-liquid pods.

ARM II: Patients receive usual care.

After completion of study intervention, patients are followed up at 2 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed lung cancer subjects will be stages I-III non-small cell lung cancer (NSCLC) and head and neck cancer subjects will be stages I-IV squamous cell carcinoma (SCC).
* Current smokers of combustible cigarettes who smoke >= 4 days/week.
* Lung cancer patients planning to undergo wedge resection surgery for their index cancer.
* Head and neck cancer patients planning to undergo surgical resection of their index cancer or exploratory biopsies (tonsil cancer).
* Patients must intend to receive ongoing oncology care at Ohio State University [OSU] (i.e., their clinic visit is not a consultation/second opinion).
* Patients that are over the age of 21 years.

Exclusion Criteria:

* Patients who are cognitively unable to understand the consent form or participate in interviews.
* Patients with hearing impairments.
* Patients who are planning to use or are currently using cessation medication to help quit or reduce smoking.
* Patients who are currently using e-cigarettes.
* Patients undergoing surgery including lobectomy, pneumonectomy, tracheotomy, laryngectomy, or free flap surgery.
* Patients with contraindications to per oral intake.
* Lung cancer patients who are on home supplemental oxygen at baseline.
* Patients that have problems with dexterity that would impact electronic cigarette use.
* Patients under 21 years of age.
* Patients who don't speak and read English.
* Patients with histologies other than NSCLC, or squamous cell carcinoma of the head and neck.
* Patients with nasopharyngeal, thyroid, or gland cancers.
* Patients with inoperable tumors.
* Pregnant women.
* Prisoners.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of patients measured by number of screened per month | Up to 6 months
  Will be measured by the number of screened patients per month.
Feasibility of patients measured by number of screened per month by eligibility status | Up to 6 months
  Will be measured by the number of screened patients per month by eligibility status.
Feasibility of patients measured by number of screened per month by refusal status | Up to 6 months
  Will be measured by the number of screened patients per month by refusal status.
Reasons for participant ineligibility | Baseline
  We will record reasons for patient ineligibility
Reasons for participant refusal | Baseline
  We will record reasons for patient refusal to participate
Acceptance measured by participation rate | Up to 6 months
  Will be measured by the participation rate, the number of eligible participants who consent and agree to study participation.
Compliance | Up to 6 months
  Will be self-reported and include counting of used JUUL pods on follow-ups interviews.
Adherence | Baseline and hospital admission for surgery
  Further, exhaled carbon monoxide (a marker of short-term smoking status) will be assessed at baseline and upon hospital admission for surgery.
Incidence of adverse events (AEs) | Up to 14 days after delivery of intervention
  Will be assessed at days 2 and 14 following the delivery of the intervention and reported by participants. Further, participants will be invited to contact the research team to report any adverse events related to the use of the intervention at any time point.
Complication rate (primary preliminary efficacy) | Up to 6 months
  Will be measured as the number of complications reported, per person month of follow up.
Quality of life (QOL) - anxiety & depression | Up to 6 months
  Self-reported QOL measures will include the GAD-7 (anxiety and depressive symptoms)
Quality of life (QOL) - anxiety & depression 2 | Up to 6 months
  Self-reported QOL measures will include the PHQ-9 (anxiety and depressive symptoms)
Quality of life (QOL) - Perceptions of cancer | Up to 6 months
  Self-reported QOL measures will include the Perceptions of Lung Cancer to assess views on their disease (modified slightly for head and neck cancer patients)
Quality of life (QOL) - Health outcomes | Up to 6 months
  Self-reported QOL measures will include the EQ-5D-5L to assess overall and cancer-specific health outcomes (including cough, dyspnea, dysphagia, and pain).
Quality of life (QOL) - Health outcomes 2 | Up to 6 months
  Self-reported QOL measures will include the and EORTC-QLQ-LC13 to assess overall and cancer-specific health outcomes (including cough, dyspnes, dysphagia, and pain).
7 day point prevalence of tobacco use | Up to 6 months
  7-day point prevalence of tobacco use (i.e., switching) will be measured at follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Brasky, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu